CLINICAL TRIAL: NCT02960256
Title: The Impact of Infectious Disease on QT Segment
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Lee Goldstein, Principal Investigator, HaEmek Medical Center, Israel
Other Study IDs: 112-16
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Sepsis; Pneumonia; Cardiomyopathy, Secondary
MeSH Terms: conditions — Sepsis; Pneumonia; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients admitted to an internal medicine department due to an
  Interventions: Device: ekocardiogram test

INTERVENTIONS:
Device: ekocardiogram test — ekocardiogram test

SUMMARY:
Sepsis related to the development of cardiac complications. However, the investigators understanding regarding this condition remains incomplete. Possible explanations raised include coronary perfusion decrease, activation of the coagulation system and release of inflammatory mediators, including endotoxins, cytokines and others.

In this study the investigators wanted to examine the impact of any infectious disease, (not necessarily Pneumonia), on the QT interval in patients hospitalized for acute infectious disease.

ELIGIBILITY:
Inclusion Criteria:

* Internal ward hospitalized patient, due to illness which its etiology is bacterial, fungal or viral

Exclusion Criteria:

* Can not technically perform reliably ECG (amputated legs, lack of cooperation, etc.)
* Subject with permanent pacemaker

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to an internal medicine department due to an infectious disease.
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Prolongation of the QT | 5 days
  QT will be measured by ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No